CLINICAL TRIAL: NCT04461938
Title: Characterization of Metabolic Changes in the Glioma Tumor Tissue Induced by Transient Fasting (ERGO3)
Acronym: ERGO3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Michael Ronellenfitsch, Princial Investigator, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ERGO3
Record Dates: First submitted 2020-03-23; First posted 2020-07-08 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Glioma, Mixed
Keywords: metabolism-nutritional intervention-ketogenic diet-fasting
MeSH Terms: conditions — Glioma | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting (Other): All study participants follow the same dietary intervention; thus, no randomization will take place.
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — The study intervention consists of one fasting cycle of 72 hours prior to biopsy/resection. Depending on clinical condition, patients can be hospitalized during the course of the study (e.g. need for medical assistance due to immobilization). Patients in good clinical condition will be admitted on day 3.

SUMMARY:
Nutritional interventions such as ketogenic diet (KD) or fasting are currently under evaluation as anti-cancer treatment. In glioma patient cohorts, the feasibility and safety of fasting in addition to antitumor treatment has been shown. However, it is still unclear whether fasting exerts effects on the glioma tumor tissue at all, and whether fasting causes metabolic or immunological changes in the glioma microenvironment that could be exploited therapeutically. Therefore, the central contribution of this study is to characterize metabolic and immunological changes in the glioma tumor tissue induced by a fasting cycle of 72 hours prior to biopsy or resection.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of glioma World Health Organization (WHO) grade II, III or IV as assessed by cerebral imaging (MRI)
* MRI-suspected relapse of previously diagnosed glioma
* interdisciplinary recommendation for resection or biopsy
* karnofsky performance status >= 60, Eastern Cooperative Oncology Group Performance Status (ECOG) <= 2
* creatinine <= 2,0 mg/dl, urea <= 100 mg/dl
* alanine aminotransferase (ALAT), alanine aminotransferase aspartate transaminase (ASAT) <= 7x upper normal limit
* international normalized ratio (INR) ≤ 1,5, thrombocytes > 100000/µl, leukocytes > 3000/µl

Exclusion Criteria:

* bowel obstruction, subileus
* insulin-dependent diabetes
* dexamethasone >4mg/day
* decompensated heart failure (NYHA > 2)
* myocardial infarction within the last 6 months, symptomatic atrial fibrillation
* severe acute infection or clinically relevant immunosuppression (HIV infection, granulocytopenia <1000/ µl, lymphocytopenia <500/ µl
* malnutrition, cachexia (BMI <18)
* other medical conditions that might increase the risk of the dietary intervention
* pregnancy
* uncontrolled thyroid function
* pancreatic insufficiency
* dementia or other clinically relevant alterations of the mental status which could impair the ability of the patient to apply to the diet or understand the informed consent of the study
* major contraindications to MRI scanning (e.g. presence of implanted MRI-incompatible cardiac devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in metabolism - induction of ketosis | 5 days
  The presence of ketone bodies in patient blood will be assessed by capillary sampling from a finger or an ear lobe. The presence of ketone bodies in urine will be assessed by urine test strips.
General metabolic changes | 5 days
  Main target parameters of MR spectroscopic imaging are detection of intracerebral ketone bodies (acetone, acetoacetate, beta-hydroxybutyrate), changes in lactate and adenosine triphosphate / adenosine diphosphate (ATP/ADP) concentrations and changes in intracellular pH (pHi) as determined from the chemical shift difference between inorganic phosphate (Pi) and phosphocreatine (PCr). Tumor tissue and healthy appearing normal white matter of the contralateral hemisphere will be examined.
  Tumor tissue will be analysed by metabolome and proteome analysis and RNA sequencing.
  Patient serum will be analysed by proteome analysis.
Immunological changes | 5 days
  Flow cytometry including T- and B-lymphocytes natural killer (NK) cells in blood samples.
  Analysis of gut microbiome prior to and following fasting.
Alterations in electric brain activity | 5 days
  Non-invasive electroencephalography (EEG) will be performed prior to and following fasting. It will be assessed with regard to chief frequencies and the presence of epilepsy-associated manifestations (e.g. epileptiform discharges, seizures).

SECONDARY OUTCOMES:
Intake of fluids and calories reported by dietary diary | 5 days
  Patients will be asked keep a dietary diary for days 0 to 4 reporting on their intake of fluids and/or calories.
Assessment to measure the tolerability of the diet by questionnaire | 5 days
  A short questionnaire of 8 aspects concerning the tolerability of the diet will be handed out. The patients will be asked to grade their consensus to each statement by 1 to 5 where "1" is defined as "not at all" and 5 as "very relevant" for daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Ronellenfitsch, Prof. Dr. Dr., Principal Investigator — Goethe University
Locations (1):
- Dr. Senckenberg Institute of Neurooncology, University Medicine Fankfurt, Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Result] Alcicek S, Dive I, Thomas DC, Prinz V, Forster MT, Czabanka M, Weber KJ, Steinbach JP, Ronellenfitsch MW, Hattingen E, Pilatus U, Wenger KJ. 2D 1H sLASER Long-TE and 3D 31P Chemical Shift Imaging at 3 T for Monitoring Fasting-Induced Changes in Brain Tumor Tissue. J Magn Reson Imaging. 2025 Jan;61(1):426-438. doi: 10.1002/jmri.29422. Epub 2024 May 9. PMID 38722043